CLINICAL TRIAL: NCT05301140
Title: Vivistim Registry for Paired VNS Therapy (GRASP)
Acronym: GRASP
Status: Recruiting | Type: Observational
Sponsor: MicroTransponder Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MT-St-REG or GRASP Registry
Record Dates: First submitted 2022-03-18; First posted 2022-03-29 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Upper Extremity Problem
Keywords: Ischemic Stroke; Paired Vagus Nerve Stimulation
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Vivistim System — VNS Paired with rehabilitation movements

SUMMARY:
The purpose of the Vivistim Registry for Paired VNS Therapy (GRASP) is to gather real-world information on patients with arm and hand deficits post-stroke who are considering Vivistim System treatment. Before and after Vivistim System implant, patient data will be collected and reported throughout the therapy process. Physicians or sites will receive appropriate remuneration for the effort and cost involved in collecting and transmitting this data to MicroTransponder Inc.

DETAILED DESCRIPTION:
The registry is a data repository of information on patients considering implant of the Vivistim System. The Vivistim System is an FDA approved (P210007) device used to help improve upper limb motor deficits after a stroke. Most patients entered into the registry will go on to be implanted with the System although those who decide not to move forward with the implant procedure can still have data collected as a non-implant comparison group (as long as either or both FM-A / WMFT assessments were collected). The primary purpose of the registry is to provide real-world usage and outcomes data on the Vivistim System. The patient outcome registry will collect acute and long-term follow-up data on Vivistim implanted patients treated with Paired Vagus Nerve Stimulation (Paired VNS™) post-FDA approval.

Historical and implant information as well as quality of life information will be gathered on patients who consider implant of the Vivistim® System. Data will be collected at baseline, 3, 6, and 12 months after implantation, as well as yearly thereafter for up to three (3) years post-implant. Patients who decide not to have the Vivistim System implanted can continue to have data collected for comparison purposes.

Contributing sites and physicians will have access to their own site data and can have anonymized summary analyses on all aggregated data; sites will not have access to other sites' individual level data. Physicians can then use the above information to facilitate patient selection and treatment. Publication (oral or written) of data in the registry, other than individual site data, will not be permitted without the express written advance approval of MicroTransponder, Inc. and the other physicians contributing to the dataset.

ELIGIBILITY:
Inclusion Criteria:

* Patients implanted with the Vivistim System for upper limb deficits associated with an ischemic stroke

Exclusion Criteria:

* Not eligible for surgery

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ischemic stroke patients implanted with the Vivistim System
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Fugl Meyer Assessment (FM-A) | 6 months
  Change in Fugl Meyer Assessment score
Wolf Motor Function Test (WMFT) | 6 months
  Change in Wolf Motor Function Test score

SECONDARY OUTCOMES:
Stroke Impact Scale (SIS) | 6 months
  Change in Stroke Impact Scale
Motor Activity Log (MAL) | 6 months
  Change in Motor Activity Log

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Mt. Sinai, New York, New York
  - Thomas Jefferson, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dawson J, Liu CY, Francisco GE, Cramer SC, Wolf SL, Dixit A, Alexander J, Ali R, Brown BL, Feng W, DeMark L, Hochberg LR, Kautz SA, Majid A, O'Dell MW, Pierce D, Prudente CN, Redgrave J, Turner DL, Engineer ND, Kimberley TJ. Vagus nerve stimulation paired with rehabilitation for upper limb motor function after ischaemic stroke (VNS-REHAB): a randomised, blinded, pivotal, device trial. Lancet. 2021 Apr 24;397(10284):1545-1553. doi: 10.1016/S0140-6736(21)00475-X. PMID 33894832
- [Background] Kimberley TJ, Pierce D, Prudente CN, Francisco GE, Yozbatiran N, Smith P, Tarver B, Engineer ND, Alexander Dickie D, Kline DK, Wigginton JG, Cramer SC, Dawson J. Vagus Nerve Stimulation Paired With Upper Limb Rehabilitation After Chronic Stroke. Stroke. 2018 Nov;49(11):2789-2792. doi: 10.1161/STROKEAHA.118.022279. PMID 30355189
- [Background] Engineer ND, Kimberley TJ, Prudente CN, Dawson J, Tarver WB, Hays SA. Targeted Vagus Nerve Stimulation for Rehabilitation After Stroke. Front Neurosci. 2019 Mar 29;13:280. doi: 10.3389/fnins.2019.00280. eCollection 2019. PMID 30983963
- [Background] Dawson J, Engineer ND, Prudente CN, Pierce D, Francisco G, Yozbatiran N, Tarver WB, Casavant R, Kline DK, Cramer SC, Van de Winckel A, Kimberley TJ. Vagus Nerve Stimulation Paired With Upper-Limb Rehabilitation After Stroke: One-Year Follow-up. Neurorehabil Neural Repair. 2020 Jul;34(7):609-615. doi: 10.1177/1545968320924361. Epub 2020 Jun 1. PMID 32476617
- [Background] Dawson J, Pierce D, Dixit A, Kimberley TJ, Robertson M, Tarver B, Hilmi O, McLean J, Forbes K, Kilgard MP, Rennaker RL, Cramer SC, Walters M, Engineer N. Safety, Feasibility, and Efficacy of Vagus Nerve Stimulation Paired With Upper-Limb Rehabilitation After Ischemic Stroke. Stroke. 2016 Jan;47(1):143-50. doi: 10.1161/STROKEAHA.115.010477. Epub 2015 Dec 8. PMID 26645257